CLINICAL TRIAL: NCT03533127
Title: A Phase III Study Comparing Efficacy and Safety of LY01008 and Bevacizumab Combined With Paclitaxel and Carboplatin for Treatment of Naïve Subjects With Metastatic or Recurrent Nonsquamous Non-small Cell Lung Cancer
Brief Title: A Study of LY01008 and Bevacizumab Combined With Paclitaxel and Carboplatin for Treatment of Naïve Subjects With Metastatic or Recurrent Nonsquamous Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LY01008
Record Dates: First submitted 2018-05-10; First posted 2018-05-22 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Non Small Cell Lung Cancer; Non Small Cell Lung Cancer Metastatic; Non Small Cell Lung Cancer Recurrent
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: The subjects will receive the treatment with LY01008 or bevacizumab combined with paclitaxel and carboplatin for 4-6 cycles, and then both groups of subjects will receive the maintenance monotherapy with LY01008
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY01008+Carboplatin/Paclitaxel (Experimental): Drug: LY01008 15 mg/kg IV every 3 weeks on Day 1 Drug: Carboplatin Carboplatin AUC 6 IV every 3 weeks on Day 1 for 4-6 cycles Drug: Paclitaxel Paclitaxel 175 mg/m2 IV every 3 weeks on Day 1 for 4-6 cycles
  Interventions: Drug: LY01008
- Bevacizumab + Carboplatin/Paclitaxel (Experimental): Drug: Bevacizumab Bevacizumab 15 mg/kg IV every 3 weeks on Day 1 Drug: Carboplatin Carboplatin AUC 6 IV every 3 weeks on Day 1 for 4-6 cycles Drug: Paclitaxel Paclitaxel 175 mg/m2 IV every 3 weeks on Day 1 for 4-6 cycles
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: LY01008 — LY01008+Carboplatin/Paclitaxel
  Arms: LY01008+Carboplatin/Paclitaxel
Drug: Bevacizumab — Bevacizumab + Carboplatin/Paclitaxel
  Arms: Bevacizumab + Carboplatin/Paclitaxel

SUMMARY:
This is a Randomized, Double-blind, Multicenter Phase III Study Comparing Efficacy and Safety of LY01008 (Recombinant Humanized Anti-Human Vascular Endothelial Growth Factor Monoclonal Antibody Injection) and Bevacizumab Combined with Paclitaxel and Carboplatin for Treatment of Naïve Subjects with Metastatic or Recurrent Nonsquamous Non-small Cell Lung Cancer

DETAILED DESCRIPTION:
The objectives are to compare the efficacy, safety and immunogenicity of LY01008 and bevacizumab combined with paclitaxel and carboplatin for treatment of subjects with metastatic or recurrent nonsquamous non-small cell lung cancer.

The subjects will receive the treatment with LY01008 or bevacizumab combined with paclitaxel and carboplatin for 4-6 cycles, and then both groups of subjects will receive the maintenance monotherapy with LY01008 until occurrence of progressive disease (PD), intolerable toxicity reaction, withdrawal of informed consent, loss to follow-up, death, conduct of other antineoplastic therapy or completion of the whole study. The doses of LY01008 and bevacizumab are 15 mg/kg in combination therapy. The dose of LY01008 in maintenance monotherapy is 15 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

* The subject has voluntarily signed the written informed consent form (ICF)
* Male or female patients aged 18 to 75 years (18 years and 75 years are inclusive)
* The patients with metastatic (stage IV) or recurrent nonsquamous NSCLC proved by histological or cytological demonstrated who cannot have surgical treatment. The diagnosis result of nonsquamous NSCLC obtained only based on the sputum cytology is not accepted. If the patient has many kinds of tumor components, the main cell types should be classified；
* The patient should have at least one measurable lesion as the target lesion (according to RECIST 1.1 criteria)；
* The Eastern Cooperative Oncology Group (ECOG) performance status score is 0 to 1 point.
* The predictable survival duration is ≥ 6 months
* Laboratory results during screening:
* Blood routine: white blood cell count ≥ 3.0× 109/L, absolute neutrophil count ≥ 1.5× 109/L, platelet count≥ 100× 109/L and hemoglobin≥ 90 g/L.
* Liver function: Total bilirubin <1.5×upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5×ULN for the subjects without liver metastasis and ALT and AST< 5×ULN for the subjects with liver metastasis.
* Kidney function: Serum creatinine ≤ 1.5 ×ULN or creatinine clearance rate ≥ 50 mL/min and urine protein <2+ ( quantitative test for 24h urine protein should be conducted when the baseline urine protein is 2+ and the subject can only be enrolled when the 24 h urine protein quantitation is ≤ 1 g );
* The international normalized ratio (INR) ≤ 1.5 and partial thromboplastin time (PTT or aPTT) ≤ 1.5 × ULN within 7 days before the study treatment
* The subject can comply with the study protocol.
* The female subjects and male subjects of childbearing age and the partners of the male subjects agree to take reliable contraceptive measures (such as abstinence, sterilizing operation, contraceptives, injection of the contraceptive drug medroxyprogesterone acetate or subdermal implant of contraceptives

Exclusion Criteria:

* The patients who have received chemotherapy or other systemic antineoplastic therapy drugs (such monoclonal antibodies and tyrosine kinase inhibitors) for the disease of the current stage (stage IV or recurrent disease). The patients are allowed to have received past surgery and radiotherapy, but they must meet the criteria for the related two treatment methods listed in the study protocol. The subjects who have recurrented after adjuvant/ neoadjuvant chemotherapy can also be enrolled if the interval between the completion time of the adjuvant/ neoadjuvant therapy and the administration time of the initial dose of the study is more than 6 months；
* The subjects with mixed NSCLC which containing small cell cancer component or the squamous-cell carcinoma component dominant；
* The patient has history of hemoptysis within 3 months before screening and the expectorated fresh blood is ≥ 2.5 mL.
* The images reveal sign of tumor invasion in great vessels. The subjects with tumor completely closes to, surrounds or invades the lumen of great vessels (such as pulmonary artery or superior vena cava) must be excluded;
* The subjects with symptomatic brain metastasis, a history of spinal cord compression or meningeal metastases and subjects who have previously received brain metastasis treatment, if their lesion is radiographically confirmed to have remained stable for more than 4 weeks at screening, can be enrolled；
* The subjects who have received radical thoracic radiotherapy within 28 days before enrollment and the subjects who have received palliative radiotherapy for the bone lesions besides chest within 2 weeks before the treatment with the first dose of study drugs；
* The subjects who have had major surgery, major trauma (such as fracture) within 28 days before randomization or the subjects who are expected to have major surgery during the study cycle ；
* The patients who are taking or have taken aspirin (>325 mg/day) or other non-steroidal anti-inflammatory drugs which are known to be able to inhibit platelet function recently (within 10 days before receiving the initial dose of the study drugs)；
* The patients who are taking or have taken whole dose oral or parenteral anticoagulation drugs or thrombolytic agents recently (within 10 days before receiving the initial dose of the study drugs). However, the patients are allowed to have preventive use of anticoagulation drugs；
* The patients who have inherited bleeding tendency or coagulation disorders；
* The patient with thrombotic diseases which revealed by medical history or examination results within 6 months before enrollment；
* The patient with uncontrolled hypertension (systolic pressure is more than 150 mmHg and/or diastolic pressure is more than 100 mmHg), hypertensive crisis or history of hypertensive encephalopathy;
* The patient with any unstable systemic disease: including but not limited to unstable angina pectoris, cerebrovascular accident or transient cerebral ischemia (within 6 months before screening), myocardial infarction (within 6 months before screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ grade II), serious arrhythmia，liver, kidney or metabolic diseases that need drug treatment,
* The patient with serious unhealed wound and gastrointestinal ulcer. Medical history of the following diseases within 6 months before screening: gastrointestinal perforation, corrosive esophagitis or gastritis, inflammatory bowel disease or diverticulitis, abdominal fistula or intra-abdominal abscess.
* The patient with tracheo-esophageal fistula；
* The patient with malignant tumors except NSCLC within 5 years before randomization, except the sufficiently treated carcinoma in situ of cervix, basal cell carcinoma or squamous epithelial cancer, local prostate cancer after radical operation, ductal carcinoma in situ after radical operation
* The patient with medical history of peripheral neuropathy;
* The patient with persistent or active infection signs which need intravenous injection of antibiotics, neurological or metabolic dysfunction, contraindications of the study drugs appear in the physical examination results or laboratory examination results or the patients have signs of suspected diseases or symptoms which result in that the patient has high risk for the treatment related complications；
* The patient with hepatitis B surface antigen (HBsAg) positive and the peripheral blood HBV DNA titer ≥1× 103 copies/mL. The subject is eligible to be enrolled if HBsAg is positive and peripheral blood HBV DNA titer <1×103 copies/mL and the investigator considers that the subject is at the stable stage of chronic hepatitis and the risk will not be increased for the subject；
* The patient with hepatitis C virus (HCV) antibody and human immunodeficiency virus (HIV) antibody positive.
* The patient has received treatment with any other investigational drugs or has participated in another interventional clinical trial within 30 days before screening
* The patient with known allergy to bevacizumab or its any excipient or paclitaxel and carboplatin drug components
* The patient has bibulosity within 1 month prior to screening (ie, drinking more than 14 units of alcohol per week (1 unit=360 mL of beer or 45 ml of 40% liquor or 150 mL of wine) or a history of drug abuse；
* Pregnant or lactating women or women who prepare to be pregnant or lactate during the study period.
* Other circumstances which are considered by the investigator that the subject is unsuitable to be enrolled

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2020-06-28 (Estimated); Study Completion 2020-12-28 (Estimated)

PRIMARY OUTCOMES:
Best Objective Response Rate | 19 weeks from randomization

SECONDARY OUTCOMES:
Progression Free Survival | from the date of randomisation to the date of disease progression or death up to 12 months from randomisation of the last subject
Overall Survival | from the date of randomisation to the date of death up to 12 months from randomisation of the last subject

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences, Chaoyang, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi Y, Lei K, Jia Y, Ni B, He Z, Bi M, Wang X, Shi J, Zhou M, Sun Q, Wang G, Chen D, Shu Y, Liu L, Guo Z, Liu Y, Yang J, Wang K, Xiao K, Wu L, Yi T, Sun D, Kang M, Ma T, Mao Y, Shi J, Tang T, Wang Y, Xing P, Lv D, Liao W, Luo Z, Wang B, Wu X, Zhu X, Han S, Guo Q, Liu R, Lu Z, Zhang J, Fang J, Hu C, Ji Y, Liu G, Lu H, Wu D, Zhang J, Zhu S, Liu Z, Qiu W, Ye F, Yu Y, Zhao Y, Zheng Q, Chen J, Pan Z, Zhang Y, Lian W, Jiang B, Qiu B, Zhang G, Zhang H, Chen Y, Chen Y, Duan H, Li M, Liu S, Ma L, Pan H, Yuan X, Yuan X, Zheng Y, Gao E, Zhao L, Wang S, Wu C. Bevacizumab biosimilar LY01008 compared with bevacizumab (Avastin) as first-line treatment for Chinese patients with unresectable, metastatic, or recurrent non-squamous non-small-cell lung cancer: A multicenter, randomized, double-blinded, phase III trial. Cancer Commun (Lond). 2021 Sep;41(9):889-903. doi: 10.1002/cac2.12179. Epub 2021 Jun 29. PMID 34184418